CLINICAL TRIAL: NCT06064214
Title: Effect of Bilateral Ultrasound-Guided Intermediate Cervical Plexus Block Combined With General Anesthesia on THE Stress Response in Patients Undergoing Anterior Cervical Spine Surgery. A Randomized Controlled Study
Brief Title: Intermediate Cervical Plexus Block on Stress Response
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed raafat taha abd el aziz, principle investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: cervical plexus block
Record Dates: First submitted 2023-09-19; First posted 2023-10-03 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Stress

STUDY DESIGN:
Intervention Model Description: randomized controlled study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- block (Experimental): 33 patients will receive bilateral u/s guided intermediate cervical plexus block with general anesthesia
  Interventions: Procedure: u/s guided intermediate cervical plexus block
- morphine (Active Comparator): 33 patients will receive morphine in a dose of 0.1-0.2 mg/kg to maintain intraoperative analgesia
  Interventions: Procedure: u/s guided intermediate cervical plexus block

INTERVENTIONS:
Procedure: u/s guided intermediate cervical plexus block — The patient will be placed in supine position,u/s probe is placed on the lateral neck, overlying the sternomastoid muscle at the level of its midpoint , Once the SCM has been identified, the transducer is moved posteriorly until the tapering posterior edge is positioned in the middle of the screen.cervical plexus is visible as a small collection of hypoechoic nodules ( immediately superficial to the prevertebral fascia the needle is passed through the skin, platysma, and investing layer of the deep cervical fascia, and the tip is placed adjacent to the plexus,bupivicaine 0.25% (5-15 mL) is administered to envelop the plexus

SUMMARY:
The aim of the present study is to investigate the effect of Bilateral Ultrasound-Guided intermediate cervical plexus Block combined with general anesthesia on the stress and inflammatory response in patients undergoing anterior cervical spine surgery (ACSS)

DETAILED DESCRIPTION:
Stress response is the name given to the hormonal and metabolic changes which follow injury or trauma. It may lead to changes in the nervous, endocrine and immune systems, and alterations in metabolic processes and functions. The stress response can shift from an adaptive and protective role to a pathogenic occurrence, especially when it is strong and chronic.

Stress hormones, the most prevalent of which is cortisol, have a circadian pattern in which they gradually climb after night sleep to reach a peak at early morning wake-up time, then gradually decline as the day progresses .

This pattern, however, can be disrupted by any stressful situation, such as severe pain from surgery, which has been linked to a progressive rise in cortisol levels both intraoperatively and in the early postoperative period.

Cytokines are group of low molecular weight proteins that modulate the systemic inflammatory response elicited by surgical intervention. Increased levels of proinflammatory cytokines, including interleukin-6 (IL-6) which is the main cytokine responsible for inducing the systemic changes, is an early features of acute injury. Interleukin-6 could be a good marker for research purposes that reflects and compares postoperative stress levels.

Spine surgeries are increasingly being performed as short-stay surgical procedures, and anterior cervical decompression and fusion is one such procedure .Postoperative incisional pain has been described as moderate in intensity, requiring opioid analgesics in most cases. Nonetheless, opioid-related side effects such as nausea, vomiting, and respiratory depression are undesirable in these patients who are at risk for airway problems due to surgical retraction or wound hematoma.

Regional anesthesia inhibits the stress response to surgery and can also influence postoperative outcomes. . The endocrinal stress response to the surgical operation is reduced as a result of inhibiting afferent impulses from the surgical site. Furthermore, a reduction in this type of stress response is seen as a key indicator of a successful regional block.

Intermediate cervical plexus block (CPB) is a safe and simple technique that has been shown to provide good pain relief through blocking all four cutaneous branches of the cervical plexus, as well as sensory and motor branches .Not only Intermediate (CPB) is superior to superficial CPB in terms of effectiveness, but also is safer than deep (CPB) .

There is a paucity of evidence for the effect of bilateral cervical plexus block for anterior cervical spine surgeries. Prior research had employed recovery questionnaire score, 24-h opioid usage and length of hospital stay in assessment of cervical plexus block effectiveness , however estimating the effect of Intermediate (CPB) on stress biomarkers as serum cortisol and interleukien-6 has not been discussed yet

ELIGIBILITY:
Inclusion Criteria:

* 1. ASA I & ASA II patients.(The American Society of Anesthesiologists) 2. Age group: from 18 to 65 years old. 3. Patients undergoing anterior cervical discectomy or fixation. 4. Genders eligible for study: both sexes

Exclusion Criteria:

* • Patient refusal.

  * Patient Undergoing posterior fixation in addition to anterior.
  * An allergy to local anaesthetics.
  * Infection at block puncture site.
  * Bleeding disorders (Coagulopathy: PTT(partial thromboplastin time) > 40seconds, INR(international normalised ratio) > 1.2, platelet count < 120 x 103 / L.).
  * Emergency surgeries & patients in sepsis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-11-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
• The serum cortisol level 24 hours postoperatively | pre operative and after 24 hours of operation
  All operations will be performed in the morning, taking into consideration circadian rhythm of hormone release. In both groups, venous blood samples to measure serum cortisol level will be collected before surgery as a baseline, then 24 hours post-operative

SECONDARY OUTCOMES:
• The serum interleukien-6 24 hours postoperatively | pre operative and after 24 hours of operation
  All operations will be performed in the morning, taking into consideration circadian rhythm of hormone release. In both groups, venous blood samples to measure serum cortisol and interleukien-6 level will be collected before surgery as a baseline, then 24 hours post-operative.interleukien-6 is normally low and may be undetectable within 30-60 min after start of surgery while reaching maximum level at 24 hours post-operative

CONTACTS AND LOCATIONS:
Overall Officials: gomaa zohry, professor, Principal Investigator — cairo universitey
Locations (1):
- Ahmed Raafat, Giza, October, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: 1 year

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-09-01): https://cdn.clinicaltrials.gov/large-docs/14/NCT06064214/Prot_SAP_000.pdf